CLINICAL TRIAL: NCT06121232
Title: Exploring the Benefit of Neuromodulation in Treating Chemo-induced Peripheral Neuropathy Using Peripheral Neuropathy Markers (Meissner's Corpuscles and Epidermal Nerve Fiber Density) and Sensory Testing (Quantitative Sensory and Gait Testing): A Single Center Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0301; NCI-2023-09269 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Neuropathy;Peripheral
MeSH Terms: conditions — Neuritis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Group 1 will receive neuromodulation.
  Interventions: Device: Abbott® DRG / Abbott®/Medtronic® SCS
- Control Group (Experimental): Group 2 will not receive neuromodulation.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Abbott® DRG / Abbott®/Medtronic® SCS — Participants will receive 1 of 2 neuromodulation procedures based on if participants are expected to have an MRI in the near future.
  Arms: Treatment Group
Other: Control Group — Participants will not receive any intervention
  Arms: Control Group

SUMMARY:
To learn if a process called neuromodulation can help to improve pain due to CIP

DETAILED DESCRIPTION:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Patients diagnosed with CIPN lower extremity due to either vinca alkaloids, taxanes, bortezomib, thalidomide, platinum-based compounds
* Patients seen at Pain Management Center at MD Anderson Cancer Center
* Patient ages greater or equal to 18 years but less than or equal to 85 years

Exclusion Criteria:

* Patients with cognitive dysfunction
* Patient with recent history (<6 months) of drug or alcohol abuse
* Patients with open skin lesion or undergoing antibiotic therapy for local for systemic infection
* Patients with painful diabetic peripheral neuropathy or preexisting peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Patients diagnosed with CIPN lower extremity due to either vinca alkaloids, taxanes, bortezomib, thalidomide, platinum-based compounds
* Patients seen at Pain Management Center at MD Anderson Cancer Center
* Patient ages greater or equal to 18 years but less than or equal to 85 years

Exclusion Criteria

* Patients with cognitive dysfunction
* Patient with recent history (<6 months) of drug or alcohol abuse
* Patients with open skin lesion or undergoing antibiotic therapy for local for systemic infection
* Patients with painful diabetic peripheral neuropathy or preexisting peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Javed, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org